CLINICAL TRIAL: NCT04915885
Title: Strengthening Contraceptive Counseling Services to Empower Clients and Meet Their Needs: Protocol for a Multi-phase Complex Intervention in Pakistan
Brief Title: Strengthening Contraceptive Counseling in Pakistan
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Additional country (Nigeria) has been added to original country, Pakistan. Therefore, an updated protocol has been submitted (NCT06081842)
Sponsor: Nguyen-Toan Tran (Other)
Responsible Party: Sponsor-Investigator, Nguyen-Toan Tran, World Health Organization consultant, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FPC21
Record Dates: First submitted 2021-05-24; First posted 2021-06-07 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Contraception
Keywords: Counseling; Empowerment; Autonomy
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (Other): routine contraceptive counseling and care and a range of family planning methods that are routinely available at field level
  Interventions: Other: Routine care
- Intervention package (Experimental): contraceptive counseling package but still with a range of family planning methods that are routinely available at field level
  Interventions: Other: Package of contraceptive counseling interventions
- Intervention package & expanded methods (Experimental): contraceptive counseling package but with an expanded range of family planning methods that are recommended by national guidance
  Interventions: Other: Package of contraceptive counseling interventions; Other: Expanded methods

INTERVENTIONS:
Other: Routine care — Routine contraceptive counseling and routine method availability
  Arms: Control arm
Other: Package of contraceptive counseling interventions — The implementation package will be co-designed by providers and clients during the formative and research design phases
  Arms: Intervention package; Intervention package & expanded methods
Other: Expanded methods — Expanded range of contraceptive methods as recommended by national policies
  Arms: Intervention package & expanded methods

SUMMARY:
High-quality contraceptive counseling can strengthen global efforts to reduce the unmet need for and suboptimal use of modern contraceptives. This study aims to identify a package of contraceptive counseling interventions designed to strengthen existing contraceptive services and determine its effectiveness in increasing clients' level of decision-making autonomy and meeting their contraceptive needs.

DETAILED DESCRIPTION:
Methods The five-phase complex intervention design starts with a pre-formative phase aimed at mapping potential study sites to establish the sampling frame. The two-part formative phase first uses participatory approaches to identify the perspectives of clients, including young people and providers, to ensure research contextualization and address each interest group's needs and priorities; clinical observations of client-provider encounters to document routine care form the second part. The design workshop of the third phase will result in the development of a package of contraceptive counseling interventions. In the fourth and experimental phase, a multi-intervention, three-arm, single-blinded, parallel cluster randomized-controlled trial will compare routine care (arm 1) with the contraceptive counseling package (arm 2) and the same package combined with wider method availability (arm 3). The fifth and reflective phase aims to analyze the package's cost-effectiveness and identify implementation barriers and enablers. The primary outcomes are clients' level of decision-making autonomy and met need for modern contraceptives.

Discussion Applying participatory action research principles in designing, testing, and scaling up effective, affordable, and sustainable counseling interventions could help optimize clients' decision-making autonomy and meet their needs for modern contraceptives in low-resource settings. Recognizing the socio-cultural and health service complexities surrounding contraception, including client-provider power dynamics, the study assumes that engaging key stakeholders, including adolescents, women, men, service providers, and policymakers would be more effective. A set of low-technology interventions will likely affect, at the individual level and in a sustainable way, the knowledge, attitudes, and behaviors of women and couples toward contraceptive counseling and provision. At the health service delivery level, the trial implementation would necessitate a shift in providers' attitudes and accountability toward a systematic integration into their clinical practice of must-have and person-centered counseling components, as well as improved health service organization to ensure the availability of competent staff and diversity of contraceptive choices.

ELIGIBILITY:
1. she comes to the family planning clinic with the intention to 1.a. use contraception for the first time in her life (new user), or 1.b. switch from a contraceptive method to another one (switching user), or 1.c. resume a method after not using any in the prior three months (lapse user), or 1.d. discontinue a modern method (discontinuing user);
2. she is not coming for the resupply of a currently used method, such as pills or injectables;
3. she has the intention to continue her follow-up at the health center during the 12-month study follow-up;
4. she does not participate in another study; and
5. she provides informed consent.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in clients' decision-making autonomy | Through study completion, an average of 1 year
  Person-Centered Contraceptive Counseling scale (PCCC), developed and tested by Dehlendorf et al. (2021)
Change in clients' met need for family planning | Through study completion, an average of 1 year
  number of participants who want to avoid a pregnancy and are using a contraceptive method / all participants

SECONDARY OUTCOMES:
Change in modern contraceptive prevalence | 6 months and 12 months post enrollment
  number of participants using a modern contraceptive / all participants

IPD SHARING:
Plan to Share IPD: Yes
(i) use of a controlled access approach, such as upon reasonable request from the World Health Organization; (ii) the trial will seek consent for sharing IPD from trial participants with adequate assurance that patient privacy and confidentiality will be maintained
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Supporting information will become available 6 months after data collection and will be available for at least 3 years
Access Criteria: Upon reasonable request from the World Health Organization